CLINICAL TRIAL: NCT00009867
Title: A PHASE II STUDY OF ARSENIC TRIOXIDE (NSC #706363, IND #57974) IN UROTHELIAL CANCER
Brief Title: Arsenic Trioxide in Treating Patients With Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02789; CALGB-99903; U10CA031946 (NIH)
Record Dates: First submitted 2001-02-02; First posted 2003-12-31 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Transitional Cell Carcinoma of the Bladder; Ureter Cancer
MeSH Terms: conditions — Urethral Neoplasms; Ureteral Neoplasms | interventions — Arsenic Trioxide

ARMS (1):
- Treatment (arsenic trioxide) (Experimental): Patients receive arsenic trioxide IV over 1 hour on days 1-5. Treatment repeats every 28 days for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response receive 2 additional courses.
  Interventions: Drug: arsenic trioxide

INTERVENTIONS:
Drug: arsenic trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid Anhydride; AS2O3; Trisenox

SUMMARY:
Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have recurrent cancer of the bladder or urinary tract. Arsenic trioxide may kill tumor cells that have become resistant to standard chemotherapy regimens.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of arsenic trioxide in patients with measurable urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis.

II. To determine the toxicity of arsenic trioxide administered to patients with urothelial cancer.

OUTLINE:

Patients receive arsenic trioxide IV over 1 hour on days 1-5. Treatment repeats every 28 days for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response receive 2 additional courses.

Patients are followed every 2 months for 1 year after registration and then every 6 months for 1 year or until disease progression or relapse.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of transitional cell carcinoma of the bladder, urethra, ureter or renal pelvis; histologic documentation of metastatic/recurrent disease is not required; clinical staging, but not pathological staging, is required
* Patients must have relapsed from or failed to achieve a complete or partial response after one chemotherapy regimen, which must have included one of the following chemotherapy agents: cisplatin, carboplatin paclitaxel, or gemcitabine
* >= 4 weeks since prior RT or chemotherapy
* Patients must have measurable disease
* CTC (ECOG) Performance Status =< 1
* No evidence of NYHA functional class III or IV heart disease
* Baseline EKG with QTc < 500 ms
* Non-pregnant and not nursing, as chemotherapy is thought to present substantial risk to the fetus/infant; men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while in this study
* Granulocytes > 1500/ml
* Platelet count > 100,000/ml
* Bilirubin =< Upper limits of normal (ULN)
* Serum Creatinine < 2.0 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-12; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Objective response | Up to 2 years
  95% confidence intervals will be computed using binomial distribution.
Toxicity graded using the CTC | Up to 2 years
  Reported by type, frequency and severity.

SECONDARY OUTCOMES:
Time to disease progression | From the initiation of treatment to the date of progressive disease, assessed up to 2 years
  Estimated using the Kaplan-Meier method.
Duration of objective response | Up to 2 years
  Estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States